CLINICAL TRIAL: NCT02748044
Title: Validation of the Utility of Rare Disease Intelligence Platform: A Multicenter Cluster Clinical Trial
Brief Title: Validation of the Utility of Rare Disease Intelligence Platform
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sun Yat-sen University (Other)
Collaborators: Ministry of Health, China (Other Government); Xidian University (Other)
Responsible Party: Principal Investigator, Erping Long, Principal Investigator, Home for Cataract Children, Zhongshan Ophthalmic Center, Sun Yat-sen University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: CCPMOH2016-China3
Record Dates: First submitted 2016-04-13; First posted 2016-04-22 (Estimated); Last update posted 2016-04-22 (Estimated); Status verified 2016-04

CONDITIONS: Cataract; Artificial Intelligence
MeSH Terms: conditions — Cataract

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Eligible patients for CC-Cruiser test (Experimental)
  Interventions: Device: CC-Cruiser

INTERVENTIONS:
Device: CC-Cruiser — An artificial intelligence to make comprehensive evaluation and treatment decision of congenital cataracts

SUMMARY:
The prevention and treatment of diseases via artificial intelligence represents an ultimate goal in computational medicine. The artificial intelligence for systematic clinical application has not yet been successfully validated. Currently, the main prevention strategy for rare diseases is to build specialized care centers. However, these centers are scattered, and their coverage is insufficient, resulting in inadequate health care among a large proportion of rare disease patients. Here, the investigators use "deep learning" to create CC-Cruiser, an intelligence agent involving three functional networks: "pick-up networks" for diagnostics, "evaluation networks" for risk stratification and "strategist networks" to provide assisted treatment decisions. The investigator also establish a cloud intelligence platform for multi-hospital collaboration and conduct clinical trial and website-based study to validate its versatility.

ELIGIBILITY:
Inclusion Criteria:

* Patients who underwent ophthalmic examination of the eye and recorded their ocular information in the collaborating hospital.

Exclusion Criteria:

-

Max Age: 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 53 (Actual)
Dates: Start 2012-01; Primary Completion 2016-04 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
The proportion of accurate, mistaken and miss detection of CC-Cruiser. | Up to 4 years

CONTACTS AND LOCATIONS:
Overall Officials: Haotian Lin, M.D., Ph.D, Study Director — Zhongshan Ophthalmic Center, Sun Yat-sen University; Yizhi Liu, M.D., Ph.D, Study Chair — Zhongshan Ophthalmic Center, Sun Yat-sen University; Erping Long, M.D., Ph.D, Principal Investigator — Zhongshan Ophthalmic Center, Sun Yat-sen University
Locations (4):
- China (4):
  - Zhongshan Ophthalmic Center, Sun Yat-sen University, Guangzhou, Guangdong
  - Department of Ophthalmology, Guangdong General Hospital, Guangdong Academy of Medical Sciences, Guangzhou, Guangdong
  - Department of Ophthalmology, First Affiliated Hospital, Guangzhou University of Traditional Chinese Medicine, Guangzhou, Guangdong
  - Department of Ophthalmology, Qingyuan People's Hospital, Qingyuan, Guangdong

REFERENCES:
- [Background] Lin H, Long E, Chen W, Liu Y. Documenting rare disease data in China. Science. 2015 Sep 4;349(6252):1064. doi: 10.1126/science.349.6252.1064-b. No abstract available. PMID 26339020
- [Background] Lin H, Ouyang H, Zhu J, Huang S, Liu Z, Chen S, Cao G, Li G, Signer RA, Xu Y, Chung C, Zhang Y, Lin D, Patel S, Wu F, Cai H, Hou J, Wen C, Jafari M, Liu X, Luo L, Zhu J, Qiu A, Hou R, Chen B, Chen J, Granet D, Heichel C, Shang F, Li X, Krawczyk M, Skowronska-Krawczyk D, Wang Y, Shi W, Chen D, Zhong Z, Zhong S, Zhang L, Chen S, Morrison SJ, Maas RL, Zhang K, Liu Y. Lens regeneration using endogenous stem cells with gain of visual function. Nature. 2016 Mar 17;531(7594):323-8. doi: 10.1038/nature17181. Epub 2016 Mar 9. PMID 26958831
- See also: Home page of Zhongshan Ophthalmic Center — http://www.gzzoc.com/
- See also: Homepage of Childhood Cataract Program of the Chinese Ministry of Health(CCPMOH) — http://www.cnccclub.com/